CLINICAL TRIAL: NCT03390894
Title: Long-Term Follow-up Study of Early Stage Breast Cancer Patients Included in GEICAM Studies
Status: Recruiting | Type: Observational
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: AECC_Asociación Española contra el Cáncer (Unknown)
Responsible Party: Sponsor
Other Study IDs: GEICAM/2016-03; 2017-002850-35 (EudraCT Number)
Record Dates: First submitted 2017-12-29; First posted 2018-01-04 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Invasive Breast Cancer Early Stages
Keywords: Long-term Follow-Up; Invasive Breast Cancer Early Stages; Previous Neoadjuvant treatment; Previous Adjuvant treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicenter, cohorts study to collect information from patients diagnosed with early-stage invasive breast cancer who have been previously included in a neoadjuvant or adjuvant clinical trial of the GEICAM group.

Patients will be included in this study from the moment of completion of the follow-up of the studies of origin and will be followed for approximately 30 years

DETAILED DESCRIPTION:
One consequence of the improvement in survival rates of certain tumors such as breast cancer is the increase in the number of patients available for long-term follow-up in randomized controlled clinical trials. This long follow-up allows an additional long-term evaluation of the efficacy, as well as of the sequelae related to the treatments that may occur beyond the time of the primary analysis.

The target population of the study are all patients who were included in neoadjuvant and adjuvant clinical trials of GEICAM performed by the goup since 1998 in the medical oncology units of the participating sites, ensuring a follow-up of patients of approximately 30 years. This will allow to describe the long-term evolution of the patients with invasive breast cancer in early stages.

The information obtained will be very useful to professionals involved in the diagnosis, treatment and monitoring of breast cancer, hospital managers, patients with this condition and society in general. This study provides data of great interest for the estimation of long-term disease requirements.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in neoadjuvant and adjuvant clinical trials with GEICAM's participation. If any of these patients had taken part or is participating in another clinical trial, she/he is eligible for this trial and her/his information will also be collected.
* Patients whose death or contact loss has not been previously collected in the databases of the original studies.

Exclusion Criteria:

* Patient who were not included in the analyses of the original studies due to non-compliance of the eligibility criteria or the original study informed consent withdrawal.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with invasive breast cancer (early stages) included in neoadjuvant and adjuvant clinical trials with GEICAM's participation.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2018-01-18 (Actual); Primary Completion 2047-01 (Estimated); Study Completion 2048-01 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival (EvFS) in neoadjuvant studies. | Throughout the whole follow up. Up to 30 years from the beginning of the Study approximately.
  The EvFS, is defined as the time from the randomization of the patients in the studies of origin, to the date of one of the following events:
  * Disease progression during neoadjuvant treatment.
  * Disease relapse (local, regional or distant) after curative surgery.
  * Second primary tumors
  * Death due to any cause.
Disease Free Survival (DFS) in adjuvant studies. | Throughout the whole follow up. Up to 30 years from the beginning of the Study approximately.
  DFS is defined as the time from the date of randomization of patients in the studies of origin, to the date of one of the following events:
  * Disease relapse (local, regional or distant) after curative surgery.
  * Second primary tumors
  * Death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS). | Throughout the whole follow up. Up to 30 years from the beginning of the Study approximately.
  Overall Survival (OS) defined as the time from the date of study enrolment to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Complejo Hospitalario de Especialidades Virgen de la Victoria; Study Director, Study Director — Hospital General Universitario Gregorio Marañón
Locations (73):
- Spain (73):
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital San Agustín Avilés, Avilés, Principality of Asturias
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Centro Oncológico de Galicia, A Coruña
  - Complejo Hospitalario A Coruña, A Coruña
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Hospital General Universitario de Alicante, Alicante
  - Hospital General Universitario de Elche, Alicante
  - Hospital General Universitario de Elda, Alicante
  - Hospital Virgen De Los Lirios, Alicante
  - Hospital Infanta Cristina, Badajoz
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Consorci Sanitari de Terrassa, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Mutua Terrassa, Barcelona
  - Instituto Catalán Oncología Barcelona Hospital Duran I Reynalds, Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Hospital Universitario de Burgos, Burgos
  - Complejo Especialidades de Jerez de la Frontera, Cadiz
  - Hospital Universitario Puerta del Mar, Cadiz
  - Complejo Hospitalario de Castellón, Castelló
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Virgen De La Luz, Cuenca
  - Hospital Universitario de Cruces, Donostia / San Sebastian
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Onkologikoa, Donostia / San Sebastian
  - Instituto Catalán de Oncología Gerona Hospital Dr. Josep Trueta, Girona
  - Hospital Universitario San Cecilio, Granada
  - Hospital Universitario Virgen De Las Nieves, Granada
  - Hospital Universitario de Guadalajara, Guadalajara
  - Complejo Hospitalario de Especialidades Juan Ramón Jiménez, Huelva
  - Complejo Hospitalario de Jaén, Jaén
  - Complejo Hospitalario Universitario de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria
  - Hospital de León, León
  - Hospital Universitario Lucus Augusti, Lugo
  - Hopsital Clínico San Carlos, Madrid
  - Hospital de Mostoles, Madrid
  - Hospital general Universitario Gregorio Marañón, Madrid
  - Hospital Madrid Montepricipe, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Fuenlabrada, Madrid
  - Hospital Universitario Fundación Alcorcón, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Severo Ochoa, Madrid
  - MD Anderson Cancer Center, Madrid
  - ALTHAIA Xarxa Asistencial Universitària Manresa, Manresa
  - Hospital Regional de Málaga Carlos Haya, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital General Universitario José María Morales Meseguer, Murcia
  - Hospital santa María Naí, Ourense
  - Complejo Hospitalario de Palencia, Palencia
  - Hospital Álvaro Cunqueiro, Pontevedra
  - Corporación Sanitaria Parc Taulí, Sabadell
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Nuestra Señora De La Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario de Valme, Seville
  - Hospital Universitario Sant Joan De Reus, Tarragona
  - Hospital Virgen de la Salud, Toledo
  - Fundación Instituto Valenciano de Oncología, Valencia
  - Hospital Arnau Vilanova, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital de Sagunto, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitari i Politécnic La Fe, Valencia
  - Hospital Universitario Dr. Peset Aleixandre, Valencia
  - Hospital de Txagorritxu, Vitoria-Gasteiz
  - Hospital Clínico Universitario de Zaragoza Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- See also: Spanish Breast Cancer Research Group (GEICAM) is a Spanish Breast Cancer Research Group — http://www.geicam.org